CLINICAL TRIAL: NCT06487416
Title: A Single-Center, Open-Label, Randomized, Single-Dose, Two-Period, Two-Sequence, Crossover Trial to Assess the Bioequivalence of Test Product Tiotropium Bromide Inhalation Powder (Strength: 18 mcg) and Reference Product (Spiriva®Handihaler®, Strength: 18 mcg) in Healthy Adult Participants Under Fasting Conditions
Brief Title: A Trial to Assess the Bioequivalence of Tiotropium Bromide Inhalation Powder in Healthy Adult Participants Under Fasting Conditions
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STXA-BE-04
Record Dates: First submitted 2024-06-28; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tiotropium Bromide Inhalation Powder (Experimental): Test Product Tiotropium Bromide Inhalation Powder (Strength: 18 microgram (mcg), as tiotropium, equivalent to 22.5 microgram of tiotropium bromide monohydrate).
  The subjects randomly received single oral dose of tiotropium bromide inhaling powder
  Interventions: Drug: Tiotropium Bromide Inhalation Powder
- Spiriva®Handihaler® (Experimental): Reference Product (Spiriva®Handihaler®, Strength: 18 microgram, as tiotropium, equivalent to 22.5 microgram of tiotropium bromide monohydrate).
  The subjects randomly received single oral dose of Spiriva®Handihaler®
  Interventions: Drug: Spiriva®Handihaler®

INTERVENTIONS:
Drug: Tiotropium Bromide Inhalation Powder — By binding to M3 receptors, the action of acetylcholine is blocked to relieve spasm of bronchial smooth muscle.
  Arms: Tiotropium Bromide Inhalation Powder
Drug: Spiriva®Handihaler® — By binding to M3 receptors, the action of acetylcholine is blocked to relieve spasm of bronchial smooth muscle.
  Arms: Spiriva®Handihaler®

SUMMARY:
Primary Objective: To evaluate the pharmacokinetics and bioequivalence of the test products Tiotropium Bromide Inhalation Powder (Strength: 18 mcg; manufactured by Chia Tai Tianqing Pharmaceutical Group Co., Ltd.) and reference products Tiotropium Bromide Inhalation Powder (Spiriva®Handihaler®, Strength: 18 mcg, manufactured by Boehringer Ingelheim Pharma GmbH and CO.KG) by oral inhalation in healthy participants under fasting conditions.

Secondary Objective: To assess the safety of the test products Tiotropium Bromide Inhalation Powder (Strength: 18 mcg) and reference products Tiotropium Bromide Inhalation Powder (Spiriva®Handihaler®, Strength: 18 mcg) in healthy participants.

ELIGIBILITY:
Inclusion Criteria:

* Able to give signed Informed Consent Form before the trial, and fully understand the trial content, process and possible adverse drug reactions (ADRs);
* Able to complete the trial in compliance with the protocol;
* Participants (including males) willing to adopt effective contraceptive methods and with no pregnancy plan from 14 days before screening to 3 months after the last scheduled visit;
* Males and females between 18 and 55 years old, inclusive;
* At least 50 kg for males, 45 kg for females, with a Body Mass Index (BMI) = Weight/Height2 (kg/m2) between 19.0-26.0 kg/m2, inclusive;
* No history of cardiac, hepatic, renal, ophthalmology and otorhinolaryngology, respiratory system, urogenital system, digestive tract, nervous system, mental and metabolic disorders, etc.

Exclusion Criteria:

* With ≥ 5 cigarettes per day on average within 3 months before screening, or not able to quit smoking during the trial, or a positive result for urine nicotine test;
* Be allergic to tiotropium, atropine or its derivatives (e.g., ipratropium, oxitropium) or any excipient of tiotropium bromide inhalation powder; or allergic constitution (be allergic to two or more drugs, food and pollen allergy); or with specific allergy history (asthma, urticaria, eczema, etc.);
* A history of alcohol abuse (alcohol consumption of more than 14 units per week: 1 unit of alcohol = 285 mL beer, or 25 mL spirits, or 100 mL wine);
* Blood donation or massive blood loss (≥400 mL) within 3 months before the initial administration; Or any blood donation plan from screening until 1 month after the last administration;
* Participants who have an acute upper respiratory tract infection within 2 weeks prior to receiving investigational product;
* History of any clinically significant diseases or any other diseases that could interfere with the study results, including but not limited to the circulatory system, gastrointestinal system, urinary system (such as history of prostate hypertrophy, bladder neck obstruction, urinary retention, etc.), respiratory system (such as acute onset of chronic obstructive pulmonary disease, pulmonary fibrosis, pulmonary hypertension, pulmonary edema, pulmonary interstitial disease, bronchospastic pulmonary disease, bronchial asthma, etc.), ophthalmology (such as: glaucoma, etc.), nervous system, immune system, endocrine system, malignant tumor, mental and metabolic abnormalities; or with history of nasopharyngitis, throat ulcers, edema, or history of throat, tracheal/bronchial and lung surgery in the past;
* Participants who have Sjogren's syndrome and habitual constipation;
* Function test: the forced expiratory volume in one second measured value / the forced expiratory volume in one second predicted value ≤80% or the forced expiratory volume in one second / forced vital capacity ≤80%;
* Any prescription medication within 14 days before the initial administration;
* Any over-the-counter (OTC) medication or Chinese herbal medicine or health supplementary within 7 days before the initial administration;
* Consumption of any special diets (such as grapefruit), or strenuous exercise engagement, or other factors affecting drug absorption, distribution, metabolism and excretion within 7 days before the initial administration;
* Participation in other drug clinical trials within 3 months before the initial administration;
* Any clinically significant abnormality findings, as judged by a clinical physician, such as physical examination, vital signs, electrocardiogram, chest X-ray examination and laboratory tests;
* Positive results of hepatitis B surface antigen, hepatitis C antibody, and HIV antibody or syphilis;
* Consumption of chocolate or any food/beverage containing caffeine or rich in xanthine within 48 h before the initial administration;
* Consumption of any products containing alcohol within 48 h before the initial administration, or a positive result of the alcohol breath test;
* A positive result of the drug abuse test, or a history of drug abuse in the past 5 years, or intake of any narcotic drugs within 3 months prior to the trial;
* A positive result of the pregnancy test, or in lactation during screening or the test period for female participants;
* History of fainting at needle or blood;
* Not tolerable on venipuncture, or a history of difficulty in venous blood collection;
* Special requirements and unable to follow the unified diet, or lactose/galactose intolerant;
* Unable to participate in this trial for participants' own reasons;
* Participants who cannot use the powder inhalers correctly after training;
* Other conditions in which participants are not suitable for the trial determined by investigators.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 186 (Actual)
Dates: Start 2024-06-10 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Peak concentration (Cmax) | Pre-dose and 1 2, 3, 4, 5 6, 7, 8, 10, 15, 20, 30 minuets, 1, 2, 4, 8, 12, 24, 48, 72, 120, 168, 216 hours post-dose
  Maximum plasma drug concentration
Area under the plasma concentration versus time curve (AUC) 0-t | Pre-dose and 1 2, 3, 4, 5 6, 7, 8, 10, 15, 20, 30 minuets, 1, 2, 4, 8, 12, 24, 48, 72, 120, 168, 216 hours post-dose
  Plasma concentration-time curve from zero to the time of the last measurable time point t
Area under the plasma concentration versus time curve (AUC) 0 - infinity | Pre-dose and 1 2, 3, 4, 5 6, 7, 8, 10, 15, 20, 30 minuets, 1, 2, 4, 8, 12, 24, 48, 72, 120, 168, 216 hours post-dose
  Area under the plasma concentration-time curve from zero to infinity

SECONDARY OUTCOMES:
The time to maximum plasma concentration (Tmax) | Pre-dose and 1 2, 3, 4, 5 6, 7, 8, 10, 15, 20, 30 minuets, 1, 2, 4, 8, 12, 24, 48, 72, 120, 168, 216 hours post-dose
  The time to maximum plasma concentration (observed)
The elimination half-life (t1/2) | Pre-dose and 1 2, 3, 4, 5 6, 7, 8, 10, 15, 20, 30 minuets, 1, 2, 4, 8, 12, 24, 48, 72, 120, 168, 216 hours post-dose
  Elimination half-life of plasma concentration
Terminal elimination rate constant (Kel) | Pre-dose and 1 2, 3, 4, 5 6, 7, 8, 10, 15, 20, 30 minuets, 1, 2, 4, 8, 12, 24, 48, 72, 120, 168, 216 hours post-dose
  Terminal elimination rate constant

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Bengbu Medical University, Bengbu, Anhui, China